CLINICAL TRIAL: NCT01281865
Title: A Phase 1b/2 Study of Imatinib in Combination With Everolimus in Synovial Sarcoma
Brief Title: Everolimus in Combination With Imatinib Mesylate in Treating Patients With Locally Advanced, Locally Recurrent, or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02577; NCI-2011-02577 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000693826; 10-167 (Other: Memorial Sloan-Kettering Cancer Center); 8603 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2013-06

CONDITIONS: Adult Synovial Sarcoma; Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma | interventions — Everolimus; Imatinib Mesylate

ARMS (1):
- Treatment (everolimus and imatinib mesylate) (Experimental): Patients receive everolimus PO once daily and imatinib mesylate PO once daily on days 1-28. Course repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood and tumor tissue sample collection at baseline and periodically during study for correlative biomarker and protein expression studies.
  Interventions: Other: diagnostic laboratory biomarker analysis; Drug: everolimus; Drug: imatinib mesylate

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis — Correlative studies
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec

SUMMARY:
This phase I/II clinical trial is studying the side effects and best dose of everolimus when given with imatinib mesylate and to see how well they work in treating patients with locally advanced, locally recurrent or metastatic soft tissue sarcoma. Everolimus and imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) of everolimus in combination with imatinib mesylate in patients with synovial sarcoma. (Phase I) II. To determine the overall response rate (RR = CR + PR). (Phase II)

SECONDARY OBJECTIVES:

I. To determine RR, progression-free survival (PFS), and overall survival (OS). (Phase I) II. To determine predictors of response. (Phase II) III. To obtain tissue biopsy and plasma samples for correlative studies pre- and post-treatment. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of everolimus followed by a phase II study.

Patients receive everolimus orally (PO) once daily and imatinib mesylate PO once daily on days 1-28. Course repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood and tumor tissue sample collection at baseline and periodically during study for correlative biomarker and protein expression studies.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed synovial sarcoma that is platelet-derived growth factor receptor, alpha polypeptide positive (PDGFRA+)
* Metastatic and/or locally advanced or locally recurrent disease
* Patients must consent to tumor biopsies before therapy and after the second week of therapy

  * Patients who do not have accessible tumor for biopsy may be enrolled at the discretion of the principal investigator
* Patients must have measurable disease, by RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan

  * Tumor lesions that are situated in a previously irradiated area may be considered measurable for the purposes of this study only if there is evidence of growth of the area following a course of irradiation that cannot be attributed to necrosis or bleeding into the tumor
* Patients with brain metastasis that has been treated with definitive surgery or radiotherapy, and who have been clinically stable for 3 months following the procedure with no neurological signs or symptoms and no requirement for systemic glucocorticoids, are eligible for study
* ECOG performance status 0-1
* Life expectancy greater than 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) (except for patients with known Gilbert syndrome)
* AST/ALT ≤ 3 times ULN
* Serum creatinine ≤ 1.5 times ULN
* Serum glucose ≤ 120 mg/dL
* Total cholesterol < 300 mg/dL
* Triglycerides < 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal, barrier method of birth control, or abstinence) during therapy and for at least 8 weeks after completion of therapy
* Patients must not have current evidence of another malignancy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus, imatinib mesylate, or other agents used in the study
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, including HIV, active hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, poorly controlled diabetes, or psychiatric illness/social situations that would limit compliance with study requirements
* No patients with significant compromised respiratory problems or an active and unexplained pneumonitis
* No concurrent combination antiretroviral therapy for HIV-positive patients
* At least 4 weeks since any number of prior chemotherapy regimens (6 weeks for carmustine or mitomycin C) for recurrent/metastatic disease

  * No prior tyrosine kinase inhibitors
* Recovered to ≤ grade 1 NCI CTCAE version 4 adverse events related to prior tumor-specific therapy
* No patients who have had major surgery within the past 4 weeks, or who have not recovered from adverse events to ≤ grade 1 NCI CTCAE adverse events associated with surgery

  * Surgical changes not expected to improve ( e.g., removal of muscle tissue) allowed
* No prior mTOR inhibitors, such as sirolimus, everolimus, ridaforolimus, or temsirolimus
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Louise Keohan, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 01/20/2011 Protocol Closed to Accrual: 10/23/2012 Primary Completion Date (if applicable):10/22/2013 Recruitment Location is the medical clinic
Groups:
- Arm 1-Treatment (Everolimus and Imatinib Mesylate): Cycle=28 days: Everolimus: 5 mg PO QD, STI571 (imatinib, Gleevec): 400 mg PO QD
- Arm 2-Treatment (Everolimus and Imatinib Mesylate): Cycle=28 days: Everolimus: 10 mg PO QD, STI571 (imatinib, Gleevec): 400 mg PO QD
Period: Overall Study
Arm/Group | Arm 1-Treatment (Everolimus and Imatinib Mesylate) | Arm 2-Treatment (Everolimus and Imatinib Mesylate)
Started | 12 | 2
Completed | 9 | 1
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1-Treatment (Everolimus and Imatinib Mesylate) | Arm 2-Treatment (Everolimus and Imatinib Mesylate) | Total
Number analyzed (Participants) | 12 | 2 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 2 | 13
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 12 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (CR + PR) Assessed by RECIST 1.1 (Phase II)
Time Frame: At 8 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1-Treatment (Everolimus and Imatinib Mesylate) | Arm 2-Treatment (Everolimus and Imatinib Mesylate)
Number analyzed (Participants) | 9 | 1
participants
  Progression of Disease | 4 | 1
  Stable Disease | 5 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1-Treatment (Everolimus and Imatinib Mesylate) | Arm 2-Treatment (Everolimus and Imatinib Mesylate)
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/2
Other Adverse Events (participants affected / at risk) | 10/12 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Treatment (Everolimus and Imatinib Mesylate) (N=12) | Arm 2-Treatment (Everolimus and Imatinib Mesylate) (N=2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Treatment (Everolimus and Imatinib Mesylate) (N=12) | Arm 2-Treatment (Everolimus and Imatinib Mesylate) (N=2)
Alanine aminotransferase increased (Investigations) | 5 (28) | 2 (4)
Alkaline phosphatase increased (Investigations) | 4 (24) | 2 (6)
Anemia (Blood and lymphatic system disorders) | 9 (57) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (19) | 2 (6)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Cholesterol high (Investigations) | 7 (45) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 3 (19) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 5 (7) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (75) | 2 (6)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 8 (48) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (27) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 5 (11) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (19) | 2 (2)
Lymphocyte count decreased (Investigations) | 4 (5) | 0 (0)
Mucositis-oral (Gastrointestinal disorders) | 4 (4) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (7) | 2 (3)
Neutrophil count decreased (Investigations) | 3 (10) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 9 (24) | 2 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Skin and subcutaneous tissue disorders Other, specify-dry split fingernails (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 8 (47) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less